CLINICAL TRIAL: NCT00927823
Title: A Phase 1, Open-Label, Dose-Escalation Study To Evaluate Safety, Pharmacokinetics, And Pharmacodynamics Of The PI3K/MTOR Inhibitor PF-04691502 In Adult Patients With Advanced Malignant Solid Tumors
Brief Title: A Trial To Assess Safety And Tolerability Of PF-04691502 In Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1271001
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — 2-amino-8-(4-(2-hydroxyethoxy)cyclohexyl)-6-(6-methoxypyridin-3-yl)-4-methylpyrido(2,3-d)pyrimidin-7(8H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04691502 Treatment (Experimental)
  Interventions: Drug: PF-04691502

INTERVENTIONS:
Drug: PF-04691502 — Once daily continuous dosing. Dose escalation to Maximally tolerated dose (MTD) until progression or discontinuation.

SUMMARY:
A phase 1 dose-escalation trial to assess the safety, tolerability, and pharmacodynamics of PF-04691502 in adult cancer patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically confirmed malignant solid tumor for which there is no currently approved treatment or which is unresponsive to currently approved therapies.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours of the first dose of PF-04961502, These patients or their partners must be surgically sterile or be postmenopausal, or must agree to use effective contraception while receiving trial treatment and for at least 3 months thereafter. Male patients or their partners must be surgically sterile or must agree to use effective contraception while receiving trial treatment and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate
* Adequate Bone Marrow Function, including:

  1. Absolute neutrophil count (ANC) ≥1500 cells/mm3
  2. Platelets ≥75,000 cells/mm3
  3. Hemoglobin ≥9 mg/dL
* Adequate Renal Function, including:

SrCr <1.5 x ULN (upper limit of normal). OR Estimated creatinine clearance ≥60 mL/min, as calculated using method standard for the institution

* Adequate Liver Function, including:

Bilirubin ≤1.5 x ULN AST (SGOT) ≤2.5 x ULN ALT (SGPT) ≤2.5 x ULN

* Adequate glucose control, including no previous diagnosis of diabetes mellitus and HbA1c <7%.
* Adequate Cardiac Function, including:

  12-Lead electrocardiogram (ECG) with normal tracing or non clinically significant changes that do not require medical intervention. QTc interval ≤470 msec and no history of Torsades des Pointes or other symptomatic QTc abnormality

Exclusion Criteria:

* Patients with known active brain metastases. Patients with previously diagnosed brain metastases are eligible if they have completed their CNS treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable
* Chemotherapy, radiotherapy (other than palliative radiotherapy to lesions that will not be followed for tumor assessment on this study, ie, non target lesions), biological or investigational agents within 2 weeks of Baseline disease assessments
* Any surgery (not including minor procedures such as lymph node biopsy) within 4 weeks of Baseline disease assessments; or not fully recovered from any side effects of previous procedures
* Prior therapy with an agent that is known or proposed to be active by action on PI3K and/or mTOR
* Prior high-dose chemotherapy requiring hematopoetic stem cell transplantation within 12 months of study treatment start
* Uncontrolled or significant cardiovascular disease:

A myocardial infarction within 12 months Uncontrolled angina within 6 months Congestive heart failure within 6 months. Diagnosed or suspected congenital long QT syndrome. Any history of ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes). Any history of second or third degree heart block (may be eligible if currently have a pacemaker) Heart rate <50/minute on pre-entry electrocardiogram Uncontrolled hypertension.

* Current use or anticipated need for food or drugs that are known potent CYP3A4 inhibitors or inducers
* Current use or anticipated need for food or drugs that are known potent CYP1A2 inhibitors or inducers
* Concurrent administration of herbal preparations
* Breast feeding: No studies have been conducted in humans to assess the impact of PF-04691502 on milk production, its presence in breast milk and its effects on the breast-fed child. Because drugs are commonly excreted in human milk and because of the potential for serious adverse reactions in nursing infants, lactating female patients are excluded from this study.
* Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drug, such as the inability to take oral medication in tablet form and malabsorption syndrome.
* Any mental disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, Buffalo, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1271001&StudyName=%20A%20Trial%20To%20Assess%20Safety%20And%20Tolerability%20Of%20PF-04691502%20In%20Cancer%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04691502 2 mg: Single oral dose of PF-04691502 2 milligram (mg) tablet in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 2 mg tablet orally once daily continuously in 21-day cycles up to 1 year unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
- PF-04691502 4 mg: Single oral dose of PF-04691502 4 mg tablet in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 4 mg tablet orally once daily continuously in 21-day cycles up to 1 year unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
- PF-04691502 8 mg: Single oral dose of PF-04691502 8 mg tablet in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 8 mg tablet orally once daily continuously in 21-day cycles up to 1 year unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
- PF-04691502 11 mg: Single oral dose of PF-04691502 11 mg tablet in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 11 mg tablet orally once daily continuously in 21-day cycles up to 1 year unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
Period: Lead-In Period
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Started | 3 | 3 | 26 | 5
Completed | 3 | 3 | 26 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Continuous Dosing Period
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Started | 3 | 3 | 26 | 5
Treated | 3 | 3 | 23 | 5
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 26 | 5
Not completed — Death | 0 | 0 | 6 | 0
Not completed — Lost to Follow-up | 1 | 1 | 9 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 2
Not completed — Other | 1 | 2 | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All participants received either PF-04691502 2 mg, 4 mg, 8 mg or 11 mg tablet as a single oral dose in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by same PF-04691502 dose orally once daily continuously in 21 day cycles up to 1 year unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after the last dose
Population: Safety analysis set included all enrolled participants who started the treatment.
Measure: Number; unit: participants
Groups:
- PF-04691502 2 mg: Single oral dose of PF-04691502 2 mg tablet in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 2 mg tablet orally once daily continuously in 21-day cycles up to 1 year unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
participants
  AEs | 3 | 3 | 25 | 5
  SAEs | 2 | 1 | 15 | 3

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was classified as per common terminology criteria for adverse events (CTCAE) version 4.0 and defined as any of the following events occurring after first dose of study medication and considered at least possibly-related to study medication. Hematological: grade 4 neutropenia (absolute neutrophil count [ANC] <500 cells per cubic millimeter [cells/mm^3]) for 1 week or greater, febrile neutropenia (fever >=38.5 degree celsius with ANC <1000/mm^3), grade 3 (50,000 cells/mm^3) and grade 4 (<25,000 cells/mm^3) thrombocytopenia; Non-Hematologic: grade 3 or 4 nausea, vomiting, or diarrhea and any clinically significant grade 3 or greater non-hematologic toxicity, despite the use of adequate/maximal medical intervention and/or prophylaxis, and any persistent, intolerable PF-04691502 related toxicity which delayed retreatment for >14 days.
Time Frame: Baseline up to Cycle 1 Day 21
Population: Safety analysis set included all enrolled participants who started the treatment.
Measure: Number; unit: participants
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
participants | 0 | 0 | 1 | 2

3. Primary Outcome: Recommended Phase-2 Dose (RP2D)
Description: RP2D was determined based on the safety profile and pharmacodynamic findings, as per investigator's discretion.
Time Frame: Baseline up to Cycle 1 Day 21
Population: Safety analysis set included all enrolled participants who started the treatment.
Measure: Number; unit: milligram
Groups:
- PF-04691502: All participants received either PF-04691502 2 mg, 4 mg, 8 mg or 11 mg tablet as a single oral dose in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by same PF-04691502 dose orally once daily continuously in 21 day cycles up to 1 year unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
Arm/Group | PF-04691502
Number analyzed (Participants) | 37
milligram | 8

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The pharmacokinetics (PK) of PF-04691502 was assessed following a single oral dose administration in lead-in-dose period (single dose PK) and repeated oral dose administration for 21 days in Cycle 1 (multiple dose PK).
Time Frame: Pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72, 96 hours post-dose in Lead-in period; pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24 hours post-dose on Cycle 1 Day 21 (C1D21)
Population: PK population included all randomized participants who received treatment and had at least 1 of the PK parameters of interest estimated. n=participants evaluable at specified time point for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
nanogram per milliliter (ng/mL)
  Single Dose: Cmax (n=3, 3, 26, 5) | 18.07 (13) | 58.29 (35) | 66.40 (41) | 82.51 (15)
  Multiple Dose: Cmax (n=3, 3, 20, 1) | 26.30 (19) | 78.91 (25) | 102.3 (41) | 89.8 (NA) — Geometric coefficient of variation was not estimable since only 1 participant was evaluable.

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: The PK of PF-04691502 was assessed following a single oral dose administration in lead-in-dose period (single dose PK) and repeated oral dose administration for 21 days in Cycle 1 (multiple dose PK).
Time Frame: Pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72, 96 hours post-dose in Lead-in period; pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24 hours post-dose on C1D21
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
hours
  Single Dose: Tmax (n=3, 3, 26, 5) | 4.00 [3.98 to 4.03] | 0.683 [0.500 to 2.02] | 2.03 [0.500 to 48.0] | 4.07 [2.02 to 8.05]
  Multiple Dose: Tmax (n=3, 3, 20, 1) | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 2.08] | 2.01 [0.500 to 6.67] | 2.15 [2.15 to 2.15]

6. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). It was evaluated following a single oral dose in lead-in-dose period (single dose PK) only.
Time Frame: Pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72, 96 hours post-dose in Lead-in period
Population: PK population included all randomized participants who received treatment and had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
ng*hr/mL | 330.3 (20) | 734.4 (18) | 1130 (41) | 1320 (32)

7. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Plasma decay half-life of PF-04691502 was assessed following a single oral dose administration in lead-in-dose period (single dose PK) and repeat oral dose administration for 21 days in Cycle 1 (multiple dose PK).
Time Frame: Pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72, 96 hours (hrs) post-dose in Lead-in period; pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24 hrs post-dose on C1D21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Groups:
- PF-04691502 2 mg: Single oral dose of PF-04691502 2 milligram (mg) tablet in lead-in period (4 to 10 days prior to Day 1) followed by PF-04691502 2 mg tablet orally, once daily, continuously in 21-day cycles up to 1 year.
- PF-04691502 4 mg: Single oral dose of PF-04691502 4 mg tablet in lead-in period (4 to 10 days prior to Day 1) followed by PF-04691502 4 mg tablet orally, once daily, continuously in 21-day cycles up to 1 year.
- PF-04691502 8 mg: Single oral dose of PF-04691502 8 mg tablet in lead-in period (4 to 10 days prior to Day 1) followed by PF-04691502 8 mg tablet orally, once daily, continuously in 21-day cycles up to 1 year.
- PF-04691502 11 mg: Single oral dose of PF-04691502 11 mg tablet in lead-in period (4 to 10 days prior to Day 1) followed by PF-04691502 11 mg tablet orally, once daily, continuously in 21-day cycles up to 1 year.
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
hours
  Single Dose: t1/2 (n=3, 3, 26, 5) | 13.23 (2.8746) | 10.87 (0.90738) | 13.77 (5.2150) | 11.66 (1.7315)
  Multiple Dose: t1/2 (n=1, 0, 5, 1) | 9.19 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 8.984 (0.70840) | 7.83 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

8. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0-∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞). It was evaluated following a single oral dose in lead-in-dose period (single dose PK) only.
Time Frame: Pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72, 96 hours post-dose in Lead-in period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
ng*hr/mL | 340.4 (18) | 741.6 (17) | 1150 (42) | 1328 (32)

9. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: AUCtau is the area under the plasma concentration time-curve from time zero to end of dosing interval (tau), where tau is the dosing interval of 24 hours. It was evaluated following repeated oral dose administration for 21 days in Cycle 1 (multiple dose PK) only.
Time Frame: Pre-dose, 30 minutes, 1, 2, 4, 6, 8, 24 hrs post-dose on C1D21
Population: PK population included all randomized participants who received treatment and had at least 1 of the PK parameters of interest estimated. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 20 | 1
ng*hr/mL | 371.7 (5) | 966.4 (25) | 1287 (46) | 1020

10. Secondary Outcome: Number of Participants With Increase From Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF)
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 2-4 minutes) were performed and average calculated. QT interval is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. QTcF is the QT interval corrected for heart rate. Corrected QT interval using Fridericia's heart rate correction formula: QTcF = QT/RR^1/3, where RR=RR interval in seconds. End of treatment (EOT) data included values from participants who came off-treatment before cycle 8.
Time Frame: Pre-dose, 30 minutes, 1, 2, 4, 8, 24, 48, hrs post-dose in Lead-in period; 1 hour post-dose on C1D8, C1D15; 1, 2, 4, 8 hours post-dose on C1D21; 1 hour post-dose C2D1, C2D15, D1 of subsequent cycles up to C8; EOT
Population: QTc analysis set included all enrolled participants who had at least 1 ECG assessment after receiving PF-04691502.
Measure: Number; unit: participants
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
participants
  Maximum QTcF Interval Increase (Change <30 msec) | 2 | 3 | 19 | 5
  MaximumQTcF Interval Increase(Change>=30to<60msec) | 1 | 0 | 7 | 0
  Maximum QTcF Interval Increase (Change >=60 sec) | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Maximum Post-dose QT Interval Corrected Using Fridericia's Formula (QTcF)
Description: as for outcome 10
Time Frame: as for outcome 10
Population: QTc analysis set included all enrolled participants had at least 1 ECG assessment after receiving PF-04691502.
Measure: Number; unit: participants
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 5
participants
  Maximum QTcF Interval (<450 msec) | 2 | 3 | 18 | 2
  Maximum QTcF Interval (450 to <480 msec) | 1 | 0 | 5 | 3
  Maximum QTcF Interval (480 to <500 msec) | 0 | 0 | 3 | 0
  Maximum QTcF Interval (>=500 msec) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Serum Glucose at Cycle 1 Day 8 (C1D8), C1D15, C2D1, C2D15, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1 and End of Treatment (EOT)
Description: Serum glucose level was measured following 4 hours fasting. EOT data included values from participants who came off-treatment before cycle 8.
Time Frame: Baseline, C1D8, C1D15, C2D1, C2D15, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1 and EOT
Population: Serum biomarker analysis set included all enrolled participants who started treatment and had baseline and on-treatment serum biomarker samples (insulin, glucose, and c-peptide) successfully analyzed for at least 1 of the biomarkers. n=participants evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 25 | 5
milligram per deciliter (mg/dL)
  Baseline (n=3, 3, 25, 5) | 87.7 (3.51) | 84.3 (0.58) | 87.3 (16.70) | 91.8 (12.44)
  Change at C1D8 (n=3, 3, 23, 5) | 14.0 (7.55) | 16.7 (27.59) | 20.0 (25.77) | 18.8 (5.26)
  Change at C1D15 (n=3, 3, 21, 3) | 16.7 (3.79) | 11.7 (19.66) | 17.0 (27.23) | 99.3 (116.43)
  Change at C2D1 (n=3, 3, 18, 1) | 8.0 (13.53) | 4.7 (14.57) | 36.8 (37.60) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Change at C2D15 (n=3, 3, 14, 1) | 12.0 (10.15) | 11.7 (16.77) | 22.6 (28.68) | 32.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Change at C3D1 (n=2, 2, 7, 0) | 39.0 (26.87) | 15.0 (28.28) | 36.0 (26.34) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C4D1 (n=2, 0, 4, 0) | 10.5 (2.12) | NA (NA) — Results not reported because none of the participants were evaluable. | 35.0 (32.38) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C5D1 (n=2, 0, 4, 0) | 21.5 (6.36) | NA (NA) — Results not reported because none of the participants were evaluable. | 71.3 (57.66) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C6D1 (n=2, 0, 4, 0) | 19.0 (4.24) | NA (NA) — Results not reported because none of the participants were evaluable. | 7.0 (41.75) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C7D1 (n=1, 0, 2, 0) | 19.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 50.5 (105.36) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C8D1 (n=1, 0, 1, 0) | 30.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 8.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at End of Treatment (n=1, 0, 17, 3) | 33.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 43.1 (94.07) | 13.7 (12.22)

13. Secondary Outcome: Change From Baseline in Serum Insulin at Cycle 1 Day 8 (C1D8), C1D15, C2D1, C2D15, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1 and End of Treatment (EOT)
Description: Serum insulin level was measured following 4 hours fasting. EOT data included values from participants who came off-treatment before cycle 8.
Time Frame: Baseline, C1D8, C1D15, C2D1, C2D15, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1 and EOT
Population: Serum biomarker analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. n=participants evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: micro International Unit/mL (mc IU/mL)
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 18 | 4
micro International Unit/mL (mc IU/mL)
  Baseline (n=3, 3, 18, 4) | 6.2 (2.67) | 5.8 (3.72) | 8.0 (5.62) | 21.4 (25.70)
  Change at C1D8 (n=3, 3, 17, 2) | 7.2 (4.17) | 38.2 (56.39) | 28.2 (27.34) | 15.4 (15.13)
  Change at C1D15 (n=3, 3, 16, 3) | 5.6 (2.32) | 8.6 (6.17) | 25.2 (33.35) | 60.5 (30.75)
  Change at C2D1 (n=2, 3, 13, 0) | 1.4 (1.08) | 11.4 (8.17) | 26.1 (17.25) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C2D15 (n=3, 3, 10, 1) | -0.1 (8.15) | 12.0 (6.64) | 12.3 (10.95) | 29.2 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Change at C3D1 (n=2, 2, 4, 0) | 36.0 (45.21) | 14.8 (16.33) | -1.0 (5.92) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C4D1 (n=1, 0, 4, 0) | 9.1 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 20.3 (15.72) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C5D1 (n=2, 0, 4, 0) | 5.7 (1.91) | NA (NA) — Results not reported because none of the participants were evaluable. | 21.2 (14.38) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C6D1 (n=1, 0, 4, 0) | 1.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 13.7 (10.53) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C7D1 (n=0, 0, 2, 0) | NA (NA) — Results not reported because none of the participants were evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 10.4 (14.71) | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at C8D1 (n=0, 0, 1, 0) | NA (NA) — Results not reported because none of the participants were evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 8.4 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable.
  Change at End of Treatment (n=1, 0, 10, 2) | 9.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Results not reported because none of the participants were evaluable. | 7.8 (14.05) | 13.1 (3.89)

14. Secondary Outcome: Change From Baseline in Serum C-peptide at Cycle 1 Day 8 (C1D8), C1D15, C2D1, C2D15, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1 and End of Treatment (EOT)
Description: Serum C-peptide level was measured following 4 hours fasting. EOT data included values from participants who came off-treatment before cycle 8.
Time Frame: Baseline, C1D8, C1D15, C2D1, C2D15, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1 and EOT
Population: Serum biomarker analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. n=participants evaluable at specified time point for each arm, respectively. Results of PF-04691502 2 mg and 4 mg arm not reported because none of the participants were evaluable.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 13 | 1
nanogram per milliliter (ng/mL)
  Baseline (n=13, 1) | 3.1 (1.79) | 3.7
  Change at C1D8 (n=13, 1) | 5.2 (3.36) | 2.0
  Change at C1D15 (n=12, 0) | 4.4 (3.58) | NA — Results not reported because none of the participants were evaluable.
  Change at C2D1 (n=10, 0) | 6.2 (3.33) | NA — Results not reported because none of the participants were evaluable.
  Change at C2D15 (n=8, 0) | 4.5 (3.62) | NA — Results not reported because none of the participants were evaluable.
  Change at C3D1 (n=3, 0) | 2.0 (1.35) | NA — Results not reported because none of the participants were evaluable.
  Change at C4D1 (n=1, 0) | 4.9 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA — Results not reported because none of the participants were evaluable.
  Change at C5D1 (n=1, 0) | 4.8 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA — Results not reported because none of the participants were evaluable.
  Change at C6D1 (n=1, 0) | 0.7 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA — Results not reported because none of the participants were evaluable.
  Change at C7D1 (n=1, 0) | 5.8 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA — Results not reported because none of the participants were evaluable.
  Change at C8D1 (n=1, 0) | 1.5 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA — Results not reported because none of the participants were evaluable.
  Change at End of Treatment (n=6, 1) | 3.4 (2.21) | 0.9

15. Secondary Outcome: Change From Baseline in Fresh Tumor Biopsy Biomarkers at Cycle 1 Day 21
Description: Fresh tumor biopsy samples analysis included assessment of status of proteins indicative of phosphoinositide 3-kinase/mammalian target of rapamycin (PI3K/mTOR) related pathways signaling status and cell cycle status. The biomarkers included phosphorylated activated kinase (AKT) S473, AKT T308, signal transducer and activator of transcription 3 (STAT3) and forkhead transcription factor Foxo1 (FKHR) T24/forkhead in rhabdomysacoma-like 1 (FKHRL1) T32. The method of analysis was reverse phase microarray (RPMA). The signal (normalized fluorescence unit [NFU]) for each pathway biomarker was normalized against the signal (NFU) for cytokeratin. The final concentration for each pathway biomarker was reported as a cytokeratin normalized fluorescence unit (NFC) value.
Time Frame: Baseline; 4 hours post-dose on C1D21
Population: Fresh tumor biopsy analysis set included all enrolled participants in the tumor biopsy cohort who started treatment and had baseline and on-treatment fresh tumor tissue successfully analyzed for at least 1 of the biomarkers. n=participants evaluable at specified time point. Only PF-04691502 8 mg treatment arm was evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: NFC
Arm/Group | PF-04691502 8 mg
Number analyzed (Participants) | 5
NFC
  Baseline: AKT S473 (n=5) | 98.5 (100.19)
  Baseline: AKT T308 (n=4) | 102.9 (61.87)
  Baseline: FKHR T24 FKHRL1 T32 (n=5) | 193.4 (120.50)
  Baseline: STAT3 (n=5) | 260.9 (192.49)
  Change at C1D21: AKT S473 (n=5) | -72.6 (82.26)
  Change at C1D21: AKT T308 (n=4) | -48.6 (40.37)
  Change at C1D21: FKHR T24 FKHRL1 T32 (n=5) | -81.5 (47.70)
  Change at C1D21: STAT3 (n=5) | -112.2 (78.14)

16. Secondary Outcome: Change From Baseline in Hair Follicle Biopsy Biomarkers at Cycle 1 Day 21
Description: Hair follicle biopsy samples analysis included assessment of status of proteins indicative of PI3K/mTOR related pathways signaling status and cell cycle status. The analytes measured were phosphorylated AKT S473, AKT T308, KI67, STAT3 (Y705) and proline-rich Akt substrate of 40 kilodaltons at Thr246 (PRAS40 T246). The method of analysis was reverse phase microarray (RPMA). The signal for each biomarker expressed as normalized fluorescence intensity (NFI) was normalized by their respective total protein concentration. This normalization was performed by dividing the biomarker NFI by total protein concentration (mg/mL) of the sample printed to give total protein normalized fluorescence unit (NFU). All clinical sample test results are reported in NFU.
Time Frame: Baseline; pre-dose, 2, 4, 24 hours post-dose on C1D21
Population: Hair follicle analysis set included participants with hair follicles collected and analyzed for biomarkers at screening and on treatment. n=participants evaluable at specified time point. Only PF-04691502 8 mg treatment arm was evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: NFU
Arm/Group | PF-04691502 8 mg
Number analyzed (Participants) | 10
NFU
  Baseline: AKT S473 (n=10) | 21.7 (10.47)
  Baseline: AKT T308 (n=7) | 50.3 (14.33)
  Baseline: KI67 (n=6) | 117.9 (41.19)
  Baseline: PRAS40 (T246) (n=7) | 136.7 (37.37)
  Baseline: STAT3 (Y705) (n=7) | 189.8 (46.52)
  Change at 0 hour: AKT S473 (n=6) | -3.0 (8.63)
  Change at 0 hour: AKT T308 (n=5) | -5.9 (12.21)
  Change at 0 hour: KI67 (n=4) | 2.0 (36.24)
  Change at 0 hour: PRAS40 (T246) (n=6) | -3.7 (39.12)
  Change at 0 hour: STAT3 (Y705) (n=4) | 2.5 (39.98)
  Change at 2 hours: AKT S473 (n=9) | -2.5 (5.47)
  Change at 2 hours: AKT T308 (n=6) | -10.9 (13.00)
  Change at 2 hours: KI67 (n=5) | -8.6 (32.67)
  Change at 2 hours: PRAS40 (T246) (n=5) | -21.2 (28.91)
  Change at 2 hours: STAT3 (Y705) (n=5) | 21.4 (62.76)
  Change at 4 hours: AKT S473 (n=7) | -2.9 (6.15)
  Change at 4 hours: AKT T308 (n=5) | 13.6 (29.98)
  Change at 4 hours: KI67 (n=3) | 27.0 (18.39)
  Change at 4 hours: PRAS40 (T246) (n=5) | -15.7 (23.74)
  Change at 4 hours: STAT3 (Y705) (n=5) | -9.3 (48.67)
  Change at 24 hours: AKT S473 (n=7) | 3.2 (9.46)
  Change at 24 hours: AKT T308 (n=3) | 7.1 (14.89)
  Change at 24 hours: KI67 (n=4) | -12.2 (31.68)
  Change at 24 hours: PRAS40 (T246) (n=6) | 10.4 (45.68)
  Change at 24 hours: STAT3 (Y705) (n=5) | -10.8 (65.89)

17. Secondary Outcome: Number of Participants With Mutation, Deletion, Amplification in Phosphatidylinositol 3-kinase (PI3K) Pathway Signaling Related Genes and/or Proteins in Biopsied Tumor Tissue
Description: Biopsied tumor tissue was analyzed for alterations in the phosphoinositide-3-kinase/rat sarcoma (PI3K/RAS) signaling pathway by molecular approaches. The biomarkers studied were phosphoinositide-3-kinase, catalytic, alpha (PIK3CA) gene mutation, PIK3CA gene amplification, and phosphatase and tensin homolog (PTEN) protein deficiency status by immunohistochemistry.
Time Frame: Baseline; 4 hours post-dose on C1D21
Population: Baseline tumor tissue biomarker analysis set: all enrolled participants who started treatment, had baseline tumor tissues (archived paraffin block/unstained slides/fresh tumor tissue) analyzed for at least 1 of biomarkers. N (number of participants analyzed)=participants evaluable for this measure. n=participants evaluable at specified time point.
Measure: Number; unit: participants
Arm/Group | PF-04691502
Number analyzed (Participants) | 18
participants
  PTEN status: Present (n=18) | 9
  PTEN status: Absent (n=18) | 9
  PIK3CA amplification: Positive (n=17) | 2
  PIK3CA amplification: Negative (n=17) | 15
  PIK3CA mutation status: Detectable (n=17) | 3
  PIK3CA mutation status: Undetectable (n=17) | 14

18. Secondary Outcome: Number of Participants With Objective Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1). Confirmed responses are those that persist on repeat imaging study >=4 weeks after initial documentation of response. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, prior to Day 1 of Cycle every odd-numbered cycle or when progressive disease was suspected
Population: Response analysis set included all participants who started treatment and had an adequate baseline tumor assessment.
Measure: Number; unit: participants
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Number analyzed (Participants) | 3 | 3 | 26 | 4
participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 13.2] | 0 [0.0 to 60.2]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04691502 2 mg | PF-04691502 4 mg | PF-04691502 8 mg | PF-04691502 11 mg
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 15/26 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 24/26 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04691502 2 mg (N=3) | PF-04691502 4 mg (N=3) | PF-04691502 8 mg (N=26) | PF-04691502 11 mg (N=5)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 5 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04691502 2 mg (N=3) | PF-04691502 4 mg (N=3) | PF-04691502 8 mg (N=26) | PF-04691502 11 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Nodal rhythm (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 8 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 15 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 8 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 3 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 17 | 4
Feeling hot (General disorders) | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 5 | 2
Oedema (General disorders) | 0 | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 4 | 0
Pain (General disorders) | 1 | 0 | 4 | 0
Pyrexia (General disorders) | 0 | 0 | 5 | 1
Thirst (General disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 11 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 10 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 4 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 5 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 3 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.